CLINICAL TRIAL: NCT01248741
Title: High Dose Rate (HDR)Prostate Brachytherapy With Vitesse tm
Brief Title: CT-validation of Ultrasound Based Planning for High Dose Rate (HDR) Prostate Brachytherapy Using Vitesse
Acronym: Vitesse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Juanita Crook, MD FRCPC, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H10-01987
Record Dates: First submitted 2010-11-03; First posted 2010-11-25 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer; Interstitial Radiation; High Dose Rate Brachytherapy; Ultrasound-based Planning Compared to CT-based Planning
Keywords: prostate cancer; interstitial radiation,; brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HDR prostate brachytherapy (Experimental): An array of 17 gauge steel needles, 20 cm in length, is inserted under Ultrasound (US) guidance into the prostate and advanced to the base of the prostate. A template is used to maintain spacing and parallelism and the needles are individually locked into the template once positioned. A continuously acquired set of US images is obtained for treatment planning purposes. Each needle is connected to a Varisource afterloader and treatment is delivered using a 10 Curie Iridium-192 source. The needles are then removed.
  Interventions: Radiation: HDR prostate brachytherapy

INTERVENTIONS:
Radiation: HDR prostate brachytherapy — HDR prostate brachytherapy to be delivered in 2 fractions of 10 Gray as a "boost" combined with external beam radiotherapy

SUMMARY:
High Dose Rate (HDR) temporary prostate brachytherapy offers a precise form of dose escalation for prostate cancer. Needles are placed, the position is confirmed and treatment is delivered. Previously High Dose Rate prostate brachytherapy was performed under TransRectal UltraSound (TRUS) guidance but planned with Computed Tomography (CT) imaging which introduced a source of error through needle displacement while transporting and repositioning patient. Recently Varian has introduced a one-step procedure where both implant and planning are based on UltraSound imaging and performed without patient repositioning. This planning system is approved by Health Canada and is commercially available.

This study will use High Dose Rate brachytherapy to treat 20 men. Treatment will be planned with TransRectal UltraSound and validated using Computed Tomography imaging.

DETAILED DESCRIPTION:
Twenty men with intermediate risk prostate cancer, suitable for the combination of external beam radiotherapy and High Dose Rate brachytherapy will be entered in this study. High Dose Rate brachytherapy will be performed using TransRectal UltraSound guidance and then planned using both cone-beam Computed Tomography and TransRectal UltraSound. Planning by Computed Tomography is to check the reliability and reproducibility of UltraSound imaging to correctly identify the needle positions. Correct needle localization is essential because this is the basis for determining source dwell positions, dose calculation and dose optimization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically proven adenocarcinoma of the prostate.
2. Patients must have intermediate risk prostate cancer. (Clinical stage ≤ T2c, Gleason score = 7 and initial prostate specific antigen (iPSA) ≤ 20, or Gleason score ≤ 6 and iPSA > 10 and ≤ 20.
3. Patients must be fit for general or spinal anaesthetic.
4. Patients must have an estimated life expectancy of at least 10 years.
5. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
6. Patients must have no contraindications to interstitial prostate brachytherapy.
7. Patients on coumadin therapy must be able to stop therapy safely for at least 7 days.

Exclusion Criteria:

* Men not able to fully understand the trial and the informed consent document
* Men suffering from claustrophobia and unable to have a Computed Tomography scan
* Men not wishing to have a cone-beam Computed Tomography scan following the insertion of the High Dose Rate brachytherapy needles to verify the accuracy of the treatment plan
* Men who cannot safely discontinue blood thinners for a few days.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Schmid, MSc, Study Director — British Columbia Cancer Agency Dept of Radiation Physics
Locations (1):
- BCCA Center for the Southern Interior, Kelowna, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 patients were recruited from the target population of men with localized prostate cancer undergoing radical radiotherapy consisting of a combination of external beam radiation and 2 fractions of 10 Gray each of High Dose Rate brachytherapy
Period: Overall Study
Arm/Group | HDR Prostate Brachytherapy
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Localized Prostate Cancer: Patients had either intermediate risk or favorable high risk disease suitable for definitive radiotherapy.
Arm/Group | Localized Prostate Cancer
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 65 [50 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 20

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Needle Tip Identification on TransRectal UltraSound Compared to Computed Tomography
Description: Precise location of the tip of each needle in 3-dimensional space relative to the prostate determines the pattern of dose delivery. Inaccuracies in needle tip location may lead to differences detected between UltraSound(US)-based and Computed Tomography (CT)-based plans.The distance of the needle tip (as identified on either CT images or US images) protruding beyond the template was measured in mm. The template acted as a fixed reference point as it was locked into the stabilizer/stepper apparatus. The 2 protrusion readings for each needle tip were compared, the difference recorded in mm, and categorized as < 1 mm, 1-2 mm, 2-3 mm and > 3 mm.
Time Frame: Treatment was planned and delivered based on ultrasound identification of needles and needle tips relative to prostate. All measurements and comparisons of measurements pertain to the day of the procedure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Localized Prostate Cancer
Number analyzed (Participants) | 20
mm | 1.1 (0.1)

ADVERSE EVENTS:
Arm/Group | Localized Prostate Cancer
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Localized Prostate Cancer (N=20)
colostomy (Gastrointestinal disorders) | 1 (1) — sigmoid stricture
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Localized Prostate Cancer (N=20)
urethral stricture (Renal and urinary disorders) | 2 (2) — urethral stricture requiring dilatation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No